CLINICAL TRIAL: NCT00802438
Title: Eosinophilic Airway Inflammation: Relationship to Remodeling and Modulation by Mepolizumab
Brief Title: Eosinophilic Airway Inflammation and Mepolizumab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-2007-0311
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-03

CONDITIONS: Asthma
Keywords: asthma; allergic inflammation; interleukin-5
MeSH Terms: conditions — Asthma | interventions — mepolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mepolizumab (Experimental): up to 3 monthly doses of 750mg i.v. mepolizumab
  Interventions: Biological: mepolizumab

INTERVENTIONS:
Biological: mepolizumab — up to three monthly doses of 750mg i.v. mepolizumab
  Other Names: anti-interleukin 5

SUMMARY:
A drug (mepolizumab) that reduces allergic inflammation will affect the function of allergy cells called eosinophils which are produced by the body in response to allergen exposure.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 18 to 50 yrs,
* History of asthma based upon presence of asthma symptoms such as cough, shortness of breath, wheeze or chest tightness,
* positive skin-prick test to a House Dust Mite extract,
* Forced expiratory volume at one second >70% predicted pre-albuterol, > 80% predicted post albuterol
* >12% increase in Forced expiratory volume at one second following inhaled albuterol (180 µg) and/or
* airway responsiveness to methacholine (PC20 <8mg/ml).
* > 20% immediate drop in FEV1 following inhaled antigen challenge.
* Safety laboratory assessments within normal ranges (labs to include complete blood count with differential, blood urea nitrogen, creatinine, aspartate aminotransferase, alanine aminotransferase, Prothrombin time, Partial Thromboplastin Time, and platelet count)
* Female subjects of child-bearing potential must have a negative urine pregnancy test (urine HCG) within 48 hours of the methacholine challenge at Visit 2 and agree to use a reliable method of birth control for the duration of the study (reliable methods of birth control can include abstinence, barrier methods, oral contraceptives, injection contraceptives or skin absorption contraceptives).
* In the opinion of the investigator, capable and willing to grant written informed consent and cooperate with study procedures and requirements.

Exclusion Criteria:

* Use of inhaled or systemic corticosteroids or leukotriene inhibitors within 1 month of screening.
* Treatment with Omalizumab (anti-IgE) within 9 months of screening visit
* Concomitant use of any other monoclonal antibody
* Respiratory infection within 4 weeks of study
* Unstable asthma as indicated by self-report of increased symptoms or increased beta-agonist use over the previous 2 weeks.
* Female subjects who are pregnant, nursing or have a pregnancy planned during the course of study
* Current smokers (defined as smoked within the last year) or a former smoker with a history of >5 pack years.
* Major health problems such as heart disease, type I and II diabetes or lung diseases other than asthma. Decisions regarding this criteria will be based upon the judgment of the investigator.
* Previous malignancy.
* Medication other than for asthma, allergies or contraception and that the investigator feels may interfere with the conduct of study (e.g. monoamine oxidase inhibitors and B-adrenergic antagonists in any form)
* Known history of allergic reaction to previous antibody administration.
* Prior treatment with an anti-interleukin-5 monoclonal antibody,
* Use of an investigational drug within 30 days of entering the study,
* History of noncompliance with medical regimens or subjects who are considered unreliable.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2008-06-01 (Actual); Primary Completion 2013-03-01 (Actual); Study Completion 2013-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nizar N Jarjour, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin- Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kelly EA, Esnault S, Liu LY, Evans MD, Johansson MW, Mathur S, Mosher DF, Denlinger LC, Jarjour NN. Mepolizumab Attenuates Airway Eosinophil Numbers, but Not Their Functional Phenotype, in Asthma. Am J Respir Crit Care Med. 2017 Dec 1;196(11):1385-1395. doi: 10.1164/rccm.201611-2234OC. PMID 28862877

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period lasted two years (July 2008 through November 2010. Participants were recruited from our Recruitment Database, through local advertisements and the local allergy/asthma clinics.
Pre-assignment Details: After a participant signs a consent form, he/she goes through an extensive screening process that includes 4 research visits to the clinic before being assigned to their treatment. The inclusion/exclusion criteria for this study was long and many subjects screen failed prior to being assigned to a treatment.
Period: Overall Study
Arm/Group | Mepolizumab
Started | 38
Completed | 10
Not Completed | 28
Not completed — Screen Failure | 20
Not completed — Withdrawal by Subject | 7
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Mepolizumab
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint of the Study is the Percent of Eosinophils in the Bronchoalveolar Lavage Fluid After Segmental Allergen Challenge, Before and After Mepolizumab Administration (Bronchoscopy #2 vs. Bronchoscopy #4).
Description: Percent of eosinophils was determined in the bronchoalveolar lavage fluid collected from the participant after segmental allergen challenge. This was done via differential cell count using Hema-3 stain. Cell differentials were determined by counting a total of 1000 cells on two cytospin preparations. The percent eosinophils were done before and after administration of mepolizumab for a specified amount of time (up to 3 months of administration).
Time Frame: before and after up to 3 months of Mepo.
Population: Participants had mild allergic asthma with a positive skin-prick test to house dust mite, ragweed, or a standardized extract of cat, a pre-180 4g albuterol FEV1 ≥70%, a post-albuterol FEV1 ≥ 80%; airway reversibility to albuterol (180 4g) ≥12% and/or airway hyper-reactivity to methacholine (PC20 ≤8 mg/ml).
Measure: Median (Inter-Quartile Range); unit: percent of bronchoalveolar eosinophils
Arm/Group | Mepolizumab
Number analyzed (Participants) | 10
percent of bronchoalveolar eosinophils
  Pre Mepolizumab | 73 [52 to 81]
  Post Mepolizumab | 31 [4 to 49]
Statistical Analysis 1: Comparison: Mepolizumab; Summaries of log-transformed data were back-transformed to the original scale and reported as geometric mean with 95% confidence interval or median within 1st and 3rd quartiles. Outcomes are summarized using least squares means with 95% confidence intervals or median with 1st and 3rd quartiles; Test type: Other; p < 0.0001, t-test, 2 sided — A two-sided p-value<0.05 was considered significant. Analyses were conducted using SAS version 9.4 (SAS Institute, Cary, NC.)

2. Secondary Outcome: Effect of Mepolizumab on Bronchoalveolar Lavage Fluid Concentrations of IL-5 Cytokine Before and After Mepolizumab
Description: IL-5 was measured via ELISA on bronchoalveolar lavage fluid before and after mepolizumab administration (up to 3 months of administration). Fluid was prepared in LowCross-Buffer to minimize potential matrix effects. A 1/2 dilution of 1X bronchoalveolar fluid was used for IL-5 detection. Data are expressed as pg/mL and are extrapolated to 1X.
Time Frame: before and after up to 3 months of Mepo
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Mepolizumab
Number analyzed (Participants) | 10
pg/ml
  Pre Mepolizumab | 409 [49 to 741]
  Post Mepolizumab | 447 [66 to 1107]
Statistical Analysis 1: Comparison: Mepolizumab; Test type: Other — Summaries of log-transformed data were back-transformed to the original scale and reported as geometric mean with 95% confidence interval or median within 1st and 3rd quartiles. Outcomes are summarized using least squares means with 95% confidence intervals or median with 1st and 3rd quartiles; p = 0.01, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Each participant was followed anywhere between 36 weeks to 45 weeks depending on treatment path.
Arm/Group | Mepolizumab
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 8/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepolizumab (N=38)
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 4 (4) — Common cold
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Back pain after a bike race
Erythema (Immune system disorders) | 1 (1) — Erythema at IV site
Pain (General disorders) | 1 (1) — Pain at IV site
Rash on neck (Skin and subcutaneous tissue disorders) | 1 (1) — Rash on neck 9 days after previous research visit - related to switching soap.
Fever (General disorders) | 1 (1) — Fever of 101.1F post bronchoscopy

LIMITATIONS AND CAVEATS:
Our small sample size limits any meaningful consideration about the mechanisms of mepolizumab's clinical action. The prolonged time commitment and inclusion of four bronchoscopies affected subject retention and limited the sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes